CLINICAL TRIAL: NCT01622959
Title: Acupuncture Versus Intravenous Morphine in the Management of Acute Pain in Emergency Department (ED)
Brief Title: Use of ACUPUNCTURE in Emergency Departement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: use of ACUPUNCTURE in ED
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Age ≥18 Years; Presigned Consentement to Participate in the Study
Keywords: emergency departement; acute pain; acupuncture; morphine
MeSH Terms: conditions — Acute Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture (Active Comparator): Inclusion criteria:
  Traumatic and non traumatic acute pain with visual analog pain scale ( VAPS) > 40 (on a scale 0-100) Age ≥18 years Presigned consentement to participate in the study.
  Exclusion criteria:
  Temperature > 37.7° C, Anticoagulation medication use or the presence of a mechanical heart valve, Skin infections that would preclude certain acupuncture points being used, Refusal, inability to consent or communication difficulties, Acute major trauma, Any form of analgesia up to 60 minutes prior to study start, An initial pain score ≤ 40 on the pain scale (score range 0-100), Opiate contraindication, Pregnancy, Presentation to the ED > 4 times in the previous 3 months with the same condition.
  Interventions: Procedure: Acupuncture
- morphine (Sham Comparator): drug:5mg of morphine followed by intravenous administration of 2,5 mg morphine each 5 min, until VAPS becomes <30%.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — -Group Acupuncture: Receiving protocol of acupuncture. Acupuncture is performed by a trained certificied resident.
  The protocols, which allow acupuncture points to be selected from a pool of pre-determined points for each condition, provide sufficient standardization to assist replication, yet are flexible enough to allow individualized treatments. These protocols also allow for additional points, such as 'ashi points', to be used at the discretion of the acupuncturist. The location of the points, angle of insertion and depth of insertion were sourced from a popular text 'A Manual of Acupuncture'.
  -Group Morphine: Receiving 5mg of morphine followed by intravenous administration of 2,5 mg morphine each 5 min, until VAPS becomes <30%. Treatment failure is defined as VAPS>30 %, 30min after beginning of the protocol. In this case, analgesic treatment was administered according to the treating physician discretion.

SUMMARY:
Pain is the most common reason that patients present to an emergency department (ED) and is often inadequately managed. Evidence suggests that acupuncture is effective for pain relief, yet it is rarely practiced in the ED.

In 1998, a United States National Institute of Health Consensus Conference Panel reviewed the status of acupuncture and concluded that: "There is sufficient evidence of acupuncture's value to expand its use into conventional medicine and to encourage further studies of its physiology and clinical value." Similarly, in 2002, the World Health Organisation (WHO) stated that acupuncture is a safe, simple and convenient therapy and that its effectiveness as analgesia has been established in controlled clinical studies.

Notwithstanding these difficulties, it has been shown that acupuncture analgesia in the treatment of chronic pain is comparable to morphine and that its better safety profile and lack of dependence makes it the preferred method of choice for these conditions.

There are very few clinical trials of acupuncture for acute pain to inform clinical practice; that's why we have the idea to do this study in our emergency department.

DETAILED DESCRIPTION:
The objective is to evaluate the efficacy and the tolerance of acupuncture compared to intravenous morphine in the management of acute pain.

The results will also identify the impact that acupuncture treatment may have upon health resource utilization in the ED setting.

It is a randomized, prospective, controlled, conducted into emergency department. Acupuncture will be applied according to Standards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA).

In all included we recorded at baseline :

Age, sex, job, comorbidity, hour of beginning of pain. Injury nature and severity assessed by the Injury Severity Score (ISS) Mechanism of the injury and radiologic findings. VAPS : 0-100%

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and non traumatic acute (<72 hours) musculoskeletal pain with visual analog pain scale ( VAS or NRS ) > 40 (on a scale 0-100)
* Age ≥18 years
* Presigned consentement to participate in the study.
* no evidence of fracture or dislocation, including ankle and knee sprains without signs of severity (ligament rupture, laxity); shoulder and elbow tendonitis; upper and lower limb mechanical pains and lower back pain with no evidence of neurological deficit; acute abdominal pain with no urgent surgical intervention including renal colic and dysmenorrhea; and acute headache .

Exclusion Criteria:

* Temperature > 37.7° C,
* Anticoagulation medication use or the presence of a mechanical heart valve,
* Skin infections that would preclude certain acupuncture points being used,
* Refusal, inability to consent or communication difficulties,
* Acute major trauma,
* Any form of analgesia up to 60 minutes prior to study start,
* An initial pain score ≤ 40 on the pain scale (score range 0-100),
* Opiate contraindication,
* Pregnancy,
* Presentation to the ED > 4 times in the previous 3 months with the same condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
analgisia effect of acupuncture | one year
  subjuctive outcome

SECONDARY OUTCOMES:
use of acupuncture in emergency departement | one year
  objective outcome

CONTACTS AND LOCATIONS:
Overall Officials: nouira semir, MD, Principal Investigator — University of Monastir
Locations (1):
- Emergency Departement, Monastir, Tunisia

REFERENCES:
- [Background] MacPherson H, White A, Cummings M, Jobst K, Rose K, Niemtzow R; STandards for Reporting Interventions in Controlled Trails of Acupuncture. Standards for reporting interventions in controlled trials of acupuncture: The STRICTA recommendations. STandards for Reporting Interventions in Controlled Trails of Acupuncture. Acupunct Med. 2002 Mar;20(1):22-5. doi: 10.1136/aim.20.1.22. PMID 11926601